CLINICAL TRIAL: NCT02951715
Title: Evaluation of the Effects of Zinc in the Management on Tinnitus Patients With Noise Induced Hearing Loss
Brief Title: Improvement of Tinnitus After Oral Zinc on Patients With Noise-induced Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Chang Gung University (Other)
Responsible Party: Principal Investigator, Chung Feng Hwang, Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102-3893A3
Record Dates: First submitted 2016-10-31; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Hearing Loss, Noise-Induced; Tinnitus, Noise Induced; Zinc Deficiency
MeSH Terms: conditions — Hearing Loss, Noise-Induced; Tinnitus | interventions — gluconic acid; Nizatidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zinc (Experimental): A full medical history assessment was performed, and each patient completed the NIHL questionnaire (Supplementary S1), audiogram, tympanogram, speech discrimination test, distortion product otoacoustic emissions (DPOAE) testing, pitch and loudness match of the tinnitus, Tinnitus Handicap Inventory (THI) and serum zinc level analyses. All tests were repeated after 2 months of treatment with zinc gluconate (Zinga 78 mg, 10 mg elemental zinc), two tablets twice per day (40 mg per day).
  Interventions: Drug: zinc gluconate

INTERVENTIONS:
Drug: zinc gluconate — 2 months of treatment with zinc gluconate (Zinga 78 mg, 10 mg elemental zinc), two tablets twice per day (40 mg per day)
  Other Names: Zinga

SUMMARY:
Twenty patients with tinnitus and a typical noise-induced hearing loss (NIHL) audiogram were included. Each subject underwent an otoscopic examination, distortion product otoacoustic emissions, tinnitus-match testing, Tinnitus Handicap Inventory (THI) and serum zinc level analyses. After 2 months of treatment with zinc, all tests were repeated.

DETAILED DESCRIPTION:
This study enrolled patients who visited our out-patient department with the primary complaint of tinnitus. A full medical history assessment was performed, and each patient underwent an otoscopic examination, a basic audiologic evaluation. We selected the patients whose audiogram data met the inclusion criteria for NIHL: 1) bilateral typical NIHL audiogram and type A tympanogram; 2) hearing threshold above 4 kilohertz (kHz) was greater than 25 dB hearing level (HL); 3) audiogram showed the characteristic 4 kHz or 6 kHz notch (average hearing threshold was 10 dB HL higher than the baseline); 4) up-turn phenomenon appeared above 6 kHz or 8 kHz, and 5) symmetrical hearing loss threshold over bilateral ears and the disparity was less than 10 dB HL. Patients with other otologic diseases were excluded.

A full medical history assessment was performed, and each patient completed the NIHL questionnaire (Supplementary S1), audiogram, tympanogram, speech discrimination test, distortion product otoacoustic emissions (DPOAE) testing, pitch and loudness match of the tinnitus, Tinnitus Handicap Inventory (THI) and serum zinc level analyses. All tests were repeated after 2 months of treatment with zinc gluconate (Zinga 78 mg, 10 mg elemental zinc), two tablets twice per day (40 mg per day).

ELIGIBILITY:
Inclusion Criteria:

* 1) bilateral typical NIHL audiogram and type A tympanogram; 2) hearing threshold above 4k Hz was greater than 25 dB HL; 3) audiogram showed the characteristic 4 kHz or 6 kHz notch (average hearing threshold was 10 dB HL higher than the baseline); 4) up-turn phenomenon appeared above 6 kHz or 8 kHz, and 5) symmetrical hearing loss threshold over bilateral ears and the disparity was less than 10 dB HL. Patients with other otologic diseases were excluded.

Exclusion Criteria:

* Patients with pregnancy, psychologic diseases and other otologic diseases were excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | 2 months
  We used the Mandarin-Chinese version of THI questionnaire to evaluate subjective tinnitus19. The severity of subjective tinnitus was divided into five subgroups including very mild (0~16 points), mild (18~36 points), moderate (38~56 points), severe (58~76 points), and very severe (78~100 points).
Serum zinc level | 2 months

SECONDARY OUTCOMES:
Pure tone audiometry (PTA) | 2 months
  Tests were conducted in a sound-treated booth (background noise level less than 30 dB A) equipped with a two-channel clinical audiometer (GSI 61).
Speech discrimination | 2 months
  Tests were conducted in a sound-treated booth (background noise level less than 30 dB A) equipped with a two-channel clinical audiometer (GSI 61).
Distortion product otoacoustic emissions (DPOAE) | 2 months
  The measurement of DPOAE used two pure-tone stimuli at frequencies of 65 dB sound pressure level (SPL) (f1) and 55 dB SPL (f2) with an f2/f1 (frequency) ratio of 1.22. The geometric mean frequencies (GM Hz) ranged from 5 to 10 kHz. The most robust DPOAE occurs at the frequency determined by the equation 2f1-f2 (recorded as DP Hz), whereas the actual cochlear frequency region assessed with DPOAE is between these two frequencies, probably close to the f2 stimulus. The stimulus intensity was defined as positive when all frequencies of 2f1-f2 tested 6 dB SPL greater than the noise floors (NF).
Pitch of tinnitus | 2 months
  When the matching procedure was first used, the level was initially set at 5 dB above the highest measured audiometric threshold (at any frequency), and the patient reported the audiometric frequency that gave the closest match to the pitch of their tinnitus, repeated three times.
Loudness of tinnitus | 2 months
  Then the level was adjusted in 2-dB steps until the patient indicated that the tone matched the loudness of their tinnitus, repeated three times.
Tinnitus loudness level (dB SL) | 2 months
  The tinnitus loudness level (dB SL) was calculated as the intensity level minus the baseline-hearing threshold

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-YEN CHIEN, Professor, Study Director — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No